CLINICAL TRIAL: NCT00425893
Title: A Randomised Controlled Trial of Face Masks and Hand Hygiene in Reducing Influenza Transmission in Households
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Peter Houck, MD, CDC
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCCID-UCI000439A; CDC Grant# 1 U01 CI000439-01
Record Dates: First submitted 2007-01-19; First posted 2007-01-23 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Influenza
Keywords: influenza; masks; transmission; hand hygiene; non-pharmacologic interventions
MeSH Terms: conditions — Influenza, Human | interventions — Hand Hygiene; Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): health education
  Interventions: Other: health education
- 2 (Experimental): hand hygiene
  Interventions: Behavioral: hand hygiene
- 3 (Experimental): masks and hand hygiene
  Interventions: Behavioral: hand hygiene; Device: face masks

INTERVENTIONS:
Behavioral: hand hygiene — alcohol-based hand wash
  Arms: 2; 3
Other: health education — Proper nutrition, etc.
  Arms: 1
Device: face masks — face masks
  Arms: 3

SUMMARY:
This study will test the effectiveness of face masks and hand cleaning in preventing the spread of influenza within households

DETAILED DESCRIPTION:
Randomised controlled trial of surgical masks and alcohol hand wash among approximately 6069 Hong Kong residents who have a household member diagnosed with influenza. Influenza in index member and secondary infection will be documented with rapid influenza tests and PCR. Minimal risk to participants.

ELIGIBILITY:
Inclusion Criteria:

* Member of family with influenza infected member

Exclusion Criteria:

* Age less than 2 yr

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6069 (Actual)
Dates: Start 2007-02; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
secondary influenza infection | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Cowling, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Cowling BJ, Chan KH, Fang VJ, Cheng CK, Fung RO, Wai W, Sin J, Seto WH, Yung R, Chu DW, Chiu BC, Lee PW, Chiu MC, Lee HC, Uyeki TM, Houck PM, Peiris JS, Leung GM. Facemasks and hand hygiene to prevent influenza transmission in households: a cluster randomized trial. Ann Intern Med. 2009 Oct 6;151(7):437-46. doi: 10.7326/0003-4819-151-7-200910060-00142. Epub 2009 Aug 3. PMID 19652172
- [Derived] Cowling BJ, Fung RO, Cheng CK, Fang VJ, Chan KH, Seto WH, Yung R, Chiu B, Lee P, Uyeki TM, Houck PM, Peiris JS, Leung GM. Preliminary findings of a randomized trial of non-pharmaceutical interventions to prevent influenza transmission in households. PLoS One. 2008 May 7;3(5):e2101. doi: 10.1371/journal.pone.0002101. PMID 18461182